CLINICAL TRIAL: NCT05753735
Title: eXtended Antibiotic Prophylaxis for Intermediate- and High-risk Glands After Pancreatoduodenectomy to Reduce Clinically Relevant PostOperative Pancreatic Fistula: A Phase 2 Randomized Control Trial (X-POPF)
Brief Title: eXtended Antibiotic Prophylaxis for Intermediate- and High-risk Glands After Pancreatoduodenectomy to Reduce CR-POPF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal investigator left the institution.
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2223
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Fistula
Keywords: Postoperative pancreatic fistula; Pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula | interventions — Piperacillin, Tazobactam Drug Combination; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, controlled, unblinded, double-arm study with 2:1 randomization to the intervention group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard perioperative antibiotics (Active Comparator): The control group will be treated according to current standard perioperative antibiotic practice, and perioperative antibiotics will not exceed 24 hours postoperatively.
  Interventions: Drug: Piperacillin/Tazobactam
- Extended antibiotic prophylaxis (Experimental): The intervention group will receive an extended duration of current standard perioperative antibiotics, then converted to amoxicillin/clavulanic at discharge
  Interventions: Drug: Piperacillin/Tazobactam; Drug: Amoxicillin/ Clavulanic acid

INTERVENTIONS:
Drug: Piperacillin/Tazobactam — Piperacillin/Tazobactam 3.375 g IV every 6 hours while inpatient following surgery, not to exceed 10 days
Drug: Amoxicillin/ Clavulanic acid — Amoxicillin/ Clavulanic acid 875/125 mg every 12 hours after discharge to complete 10 days total antibiotics
  Arms: Extended antibiotic prophylaxis

SUMMARY:
The purpose of this clinical trial is to investigate if prolonged antibiotics after pancreatoduodenectomy can prevent the development of a pancreatic fistula and related complications. Participants who are at high risk of pancreatic fistula will be administered an extended course of antibiotics. While inpatient, the patient will receive these antibiotics through the vein, and after discharge, the antibiotics will be taken by mouth.

DETAILED DESCRIPTION:
Pancreatoduodenectomy (PD) is a commonly performed surgical procedure utilized in the treatment of either localized malignancies or benign conditions that involve the pancreatic head, 2nd/3rd portions of the duodenum, ampulla of Vater, and distal biliary system. Historically, there has been little improvement in the rate of postoperative pancreatic fistula (POPF), which occurs in approximately 10-40% of patients, and is influenced by a number of factors, including surgeon experience, pancreatic gland texture, pancreatic duct size, and underlying diagnosis. POPF is the leaking of enterically contaminated and amylase-rich fluid from the pancreatic-jejunal anastomosis created during PD. This leak may lead to serious complications. The concept of antibiotic mitigation prior to development of a CR-POPF in patients at higher risk of developing CR-POPF is an option that will be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing planned, elective pancreatoduodenectomy at University Hospitals Cleveland Medical Center (UH CMC) for any indication.
* Age >18 years. Pancreatoduodenectomy is rarely, if ever performed in the elective setting for the pediatric population at UH CMC. Therefore, this study will not include this small and different population of patients undergoing pancreatoduodenectomy.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Creatinine Clearance greater than 40 ml/min

Exclusion Criteria:

* Concurrent participation in another clinical trial, where participation in the proposed clinical trial that prohibits participation in this clinical trial, or where subjects would be actively receiving another investigational agent during the 90-day evaluation period of this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Piperacillin, Tazobactam, Amoxicillin, Clavulanic Acid or other agents used in this study.
* Subjects who are found to have another active infection or presumed infection at time of surgery who will be treated per standard of care with antibiotics regardless of randomization status.
* Subjects who are found to have metastatic disease at time of planned pancreatoduodenectomy, if surgery is otherwise aborted, or if total pancreatectomy is performed due to interoperative considerations
* Any subject who, while not having history of adverse reaction to similar chemical or biologic composition to Piperacillin, Tazobactam, Amoxicillin, Clavulanic Acid or other agents used in this study, develops a suspected drug reaction to the standard perioperative dose of antibiotic, prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Ocuin, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Loftus A, Wu VS, Elshami M, Hue JJ, Ocuin LM. Hospital charge and resource use analysis of extended-spectrum penicillin antibiotic therapy after pancreatoduodenectomy in intermediate- and high-risk patients. HPB (Oxford). 2025 Jan;27(1):63-70. doi: 10.1016/j.hpb.2024.09.011. Epub 2024 Sep 28. PMID 39424467
- [Derived] Ocuin LM, Loftus A, Elshami M, Hue JJ, Musonza T, Ammori JB, Winter JM, Hardacre JM. Extended antibiotic therapy is associated with a lower rate of clinically relevant postoperative pancreatic fistula after pancreatoduodenectomy in intermediate- and high-risk patients: A single-institution analysis. Surgery. 2024 Feb;175(2):477-483. doi: 10.1016/j.surg.2023.09.049. Epub 2023 Nov 7. PMID 37940433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Started | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants analyzed in the standard perioperative antibiotic group is zero because no patients were randomized to this arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 3 | 3
  Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 2 | 2
  Unknown or Not Reported |  | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 3 | 3
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinically Relevant (Grade B/C) Postoperative Pancreatic Fistula Rate
Description: To demonstrate that extended antibiotic prophylaxis in patients with intermediate/high fistula risk score who undergo PD reduces the rate of clinically relevant postoperative pancreatic fistula in the intervention group.
Time Frame: 56 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 1

2. Secondary Outcome: Mortality
Description: Rate of mortality
Time Frame: At 30 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

3. Secondary Outcome: Mortality
Description: Rate of mortality
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

4. Secondary Outcome: Index Postoperative Length of Stay
Description: Index postoperative length of stay
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Days |  | 6.67 (1.25)

5. Secondary Outcome: Composite Length of Stay
Description: Composite 90-day length of stay
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Days |  | 21.33 (18.37)

6. Secondary Outcome: Readmission
Description: Rate of readmission
Time Frame: At 30 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Number; unit: number of readmissions
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
number of readmissions |  | 3

7. Secondary Outcome: Readmission
Description: Rate of readmission
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Number; unit: number of readmissions
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
number of readmissions |  | 7

8. Secondary Outcome: Delayed Gastric Emptying
Description: Rate of delayed gastric emptying
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

9. Secondary Outcome: Image-guided Drain Placement
Description: Rate of image-guided drain placement
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 1

10. Secondary Outcome: Postpancreatectomy Hemorrhage
Description: Presence of postpancreatectomy hemorrhage
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

11. Secondary Outcome: Superficial Surgical Site Infection
Description: Presence of superficial surgical site infection
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

12. Secondary Outcome: Deep Surgical Site Infections
Description: Presence of deep surgical site infections
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

13. Secondary Outcome: Deep Space Infections/Intra-abdominal Abscess
Description: Presence of deep space infections/intra-abdominal abscess
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 1

14. Secondary Outcome: Additional Drain Placement
Description: Rate of additional drain placement
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 1

15. Secondary Outcome: Unplanned Return to Operating Room
Description: Measuring occurrences of unplanned return to operating room
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

16. Secondary Outcome: Acute Kidney Injury
Description: Rate of the presence of acute kidney injury
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

17. Secondary Outcome: C. Difficile Colitis
Description: Rate of the presence of C. difficile colitis
Time Frame: At 90 days
Population: Zero participants were randomized to the standard perioperative antibiotic arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
Number analyzed (Participants) | 0 | 3
Participants |  | 0

ADVERSE EVENTS:
Time Frame: 120 days (from surgery through 30 days after the final dose of prophylactic antibiotic, approximately 90 days).
Description: The number of participants at risk for All-Cause Mortality is zero in the Standard Perioperative Antibiotics group because no participants were randomized to this group.
Arm/Group | Standard Perioperative Antibiotics | Extended Antibiotic Prophylaxis
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3

LIMITATIONS AND CAVEATS:
The Principal Investigator left University Hospitals Cleveland Medical Center. Therefore, this clinical trial was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT05753735/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT05753735/ICF_001.pdf